CLINICAL TRIAL: NCT01177332
Title: Effects of Acute Elevation of Circulating Fatty Acids on Hepatic Lipid Accumulation and Metabolism in Healthy Overweight and Obese Men
Brief Title: Elevated Circulating FFA and Intrahepatic Lipid Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEC 10-3-024
Record Dates: First submitted 2010-08-02; First posted 2010-08-09 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes; Hepatic Steatosis
Keywords: FFA; Liver; steatosis; exercise
MeSH Terms: conditions — Diabetes Mellitus; Fatty Liver; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted (Experimental): Two-hour cycling test, fasted condition
  Interventions: Other: exercise
- Glucose-fed (Other): Two-hour cycling test, glucose-fed condition
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — 2 hours cycling exercise at 50 % of maximal power output

SUMMARY:
There is increasing evidence that hepatic lipid content (IntraHepatic Lipid, IHL) markedly increases the risk of metabolic complications, including insulin resistance and cardiovascular events. The investigators hypothesize that the liver is passively taking up free fatty acids (FFA) when the availability is high, thereby leading to an increased storage. To test this hypothesis, the investigators want to manipulate FFA levels, by means of a fasted exercise and recovery protocol, and monitor IHL content and hepatic Adenosine triphosphate (ATP) and inorganic phosphate (Pi) concentrations.

DETAILED DESCRIPTION:
In the Netherlands and worldwide, the number of individuals suffering from type 2 diabetes mellitus is rising steadily. As a consequence, a dramatic increase in diabetes-related morbidity and mortality can be expected over the next few decades. Accordingly, a concerted effort aimed at reducing diabetes rates and towards effective diabetes management is needed.

One of the earliest hallmarks of type 2 diabetes is resistance of the peripheral tissues liver and muscle to the action of insulin, which is generally referred to as insulin resistance. Development of insulin resistance is strongly promoted by obesity. In fact obesity is the major risk factor for insulin resistance, and 80% of all type 2 diabetic patients are overweight or obese. Whereas obesity is by definition characterized by an excessive accumulation of fat in the body, it is specifically the accumulation of fat within peripheral tissues (called steatosis or ectopic fat accumulation), which is associated with the development of insulin resistance. Indeed, type 2 diabetic patients and their first-degree relatives are characterized by excessive accumulation of fat in skeletal muscle. Similarly, the presence of fatty liver in patients with type 2 diabetes and obesity has long been reported. This accumulation of fat in the liver markedly increases the risk for metabolic complications, including insulin resistance and cardiovascular events. Despite the well-known detrimental effects of ectopic fat accumulation, it is not completely understood why fat accumulates in muscle and liver.

In recent years, non-invasive methods like proton magnetic resonance spectroscopy (1H-MRS) have been developed for quantifying lipid content in skeletal muscle and the liver, and were frequently applied by us and others. These measurements can be combined with other Magnetic Resonance techniques to investigate hepatic ATP- and Pi concentrations, determined by phosphorus magnetic resonance spectroscopy (31P-MRS). Furthermore, it has been shown that ATP- and Pi concentrations are lower in subjects with type 2 diabetes mellitus, who are characterized by hepatic lipid accumulation and hepatic insulin resistance. It has been suggested that a decreased ATP and Pi concentration may be an underlying factor for hepatic lipid accumulation.

Human studies using hepatic 1H-MRS reported that intrahepatic lipid (IHL) content is associated with obesity, the metabolic syndrome and diabetes. Furthermore, a period of 36 hours of fasting increased IHL dramatically. These conditions are characterized by elevated plasma FFA levels. We hypothesize that an increased passive uptake of FFAs can lead to a mismatch between uptake and oxidation when FFA availability is high.

Interestingly, results in skeletal muscle show that elevation of FFA levels by lipid infusion result in increased lipid content after 4 hours. Similarly, we showed that skeletal muscle lipid content is increased in the inactive arm muscle after prolonged cycling exercise in the fasted state, where FFA typically increase to up to 1450 mmol. These results suggest that high circulatory FFA levels lead to unrestrained uptake of these FA in skeletal muscle, independent of oxidative needs. Whether IHL accumulation is also the resultant of elevated plasma FFA levels is currently unknown.

Please note that in the study cited above, whereas skeletal muscle lipid content increased in the inactive arm muscle, it decreased in the active vastus lateralis muscle, reflecting the use of intramuscular lipid stores as substrate during prolonged muscular activity. Whether intensified use of IHL during exercise also leads to a decrease in IHL is presently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 40-65 years
* Overweight/obese, BMI 25-35 kg/m2
* Healthy
* Stable dietary habits
* No medication use

Exclusion Criteria:

* Female sex
* Fasting plasma glucose >6.1 mmol/l
* Haemoglobin <7.8 mmol/l
* Engagement in programmed exercise > 2 hours total per week
* Elevated liver enzymes: ALAT > 45 U/L, ASAT > 35 U/L, ALP> 140 U/L, Gamma-GT > 70 U/L
* Hypertension: blood pressure > 140 mmHg systolic or 90 mmHg diastolic
* First degree relatives with history of liver disease and diabetes mellitus
* Any medical condition requiring treatment and/or medication use
* Alcohol consumption of more than 20 g per day (± 2 units)
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in another biomedical study within 1 month prior to the screening visit
* Contraindications for MRI scan

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Intrahepatic lipid content (IHL) and hepatic ATP and PI concentrations | Day 1
  After a baseline MRI/MRS-scan, subjects will cycle for two hours, immediately after cycling another MRI/MRS-scan will be performed and again four hours post exercise. The baseline and the 4-hour post exercise MRI/MRS scans take about 1.5 hour, including both determination of IHL content, by 1H-MRS, and hepatic ATP and Pi concentrations, by 31P-MRS. The MRI/MRS scan performed directly after exercise will take about 45 min, because here only the IHL content will be determined.
Intrahepatic lipid content (IHL) and hepatic ATP and PI concentrations | Day 8
  After a baseline MRI/MRS-scan, subjects will cycle for two hours, immediately after cycling another MRI/MRS-scan will be performed and again four hours post exercise. The baseline and the 4-hour post exercise MRI/MRS scans take about 1.5 hour, including both determination of IHL content, by 1H-MRS, and hepatic ATP and Pi concentrations, by 31P-MRS. The MRI/MRS scan performed directly after exercise will take about 45 min, because here only the IHL content will be determined.

SECONDARY OUTCOMES:
Substrate oxidation and blood plasma levels of FFA, triglycerides, glucose and catecholamines | Day 1
Substrate oxidation and blood plasma levels of FFA, triglycerides, glucose and catecholamines | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Doctor, Study Director
Locations (1):
- Department of Human Biology, Maastricht University, Maastricht, Netherlands